CLINICAL TRIAL: NCT02096302
Title: Evaluar el Efecto de Una fórmula Infantil Enriquecida Con el probiótico CECT7210 Sobre la Incidencia de Infecciones Gastrointestinales
Brief Title: The Effects of an Infant Formula Containing Probiotic CECT7210 on Gastrointestinal Health
Acronym: GO-INF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Ordesa (Industry)
Collaborators: Harrison Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GO-INF-010
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Gastrointestinal Diseases
Keywords: Probiotics; Infant Formula; Microbiota; Bifidobacterium longum biovar infantis CECT7210; Growth
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Formula (Experimental): Infant formula with a novel probiotic CECT7210
  Interventions: Dietary Supplement: Infant Formula with a novel probiotic CECT7210
- Standard Formula (Active Comparator): Standard infant formula without probiotics
  Interventions: Dietary Supplement: Standard formula

INTERVENTIONS:
Dietary Supplement: Infant Formula with a novel probiotic CECT7210 — Bottle-feeding with a new infant formula enriched with probiotic CECT7210 during the first 3 months of life.
  Arms: Experimental Formula
Dietary Supplement: Standard formula — Standard formula without probiotics
  Arms: Standard Formula

SUMMARY:
The purpose of this study is to determine whether an infant formula supplemented with a new probiotic CECT7210, is effective in reducing the incidence of infections, specially the gastrointestinal ones.

DETAILED DESCRIPTION:
This a multicenter, controlled, randomized, prospective, parallel, double-blinded study to evaluate the effect of an infant formula containing a new probiotic, Bifidobacterium longum biovar infantis CECT7210, on the incidence of diarrhea in healthy infants born at term. Infants will be randomized to take an standard infant formula or the infant formula with the probiotic CECT7210 during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Full-term healthy newborns (>= 37 weeks)
* Birth weight between >=2.500g and <=4.500g)
* Normal growth curve (between 3-97 percentiles)
* 0-60 days of age on enrolment
* Maximum 30 days of breastfeeding
* Exclusively infant formula on enrolment
* Breastfeeding or infant formula with pre/probiotics feeding stopped 15 days before enrolment
* Parents or caregivers agree to exclude any source of prebiotics or probiotics during the study
* Parents or caregivers agree to follow-on the study 12 weeks
* Informed consent signed ( Parent/Legal representative)

Exclusion Criteria:

* Congenital illness or malformation that may affect infant feeding and /or normal growth
* Significant pre-natal or post-natal diseases
* Infant's family history of atopy
* Any pathology related to the immune or gastrointestinal system.
* Suspected or known allergy to cow's milk protein
* Infants receiving pre or probiotics within less than 15 days prior to enrolment
* Infant's family who in the investigator's assessment cannot be expected to comply with the protocol

Max Age: 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in diarrhea incidence | At 4th, 8th, 12th weeks
  Differences between diarrhea incidence amongst groups from baseline to 12th weeks.

SECONDARY OUTCOMES:
Changes in infections incidence | At 4th, 8th, 12th weeks.
  Differences between rate of infections or duration amongst groups.
Changes in microbiota | At 4th, 8th, 12th weeks
  Differences between faecal bacterial populations.
Changes in Immunoglobulin A secretor (IgAs) | At 4th and 12th weeks
  Differences between faecal IgAs amongst groups.
Tolerability of the product | At 4th, 8th and 12th weeks
  To evaluate gastrointestinal tolerability of both study formulas.
Growth | At 4th, 8th and 12th weeks
  To compare anthropometric measurements between probiotic CECT7210 formula group and standard group.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Polanco, Professor, Study Chair — Hospital Universitario La Paz; Joaquin Escribano, Professor, Principal Investigator — Hospital Sant Joan de Reus, Reus, Spain; Ricardo Closa, Professor, Principal Investigator — Hospital Joan XXIII de Tarragona, Tarragona, Spain
Locations (3):
- Spain (3):
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital Universitario La Paz, Madrid
  - Hospital Joan XXIII, Tarragona

REFERENCES:
- [Result] Closa R, Ferré N, Luque V, Gispert-Llaurado M, Ruibio-Torrents C, Polanco I, Morera M, Moreno JA, Rivero M, Escribano J. Effect of probiotic CECT7210 supplementation of infant formula in healthy infants. ESPGHAN Abstracts Book. JPGN. Vol. 60, Supplement 1, May 2015. PA-N-0038.
- [Result] Moreno JA, Cifuentes GC, Morera M, Martínez-Blach JF, Codoñer F, Genovés S, Chenoll E, Polanco I, Closa R, Escribano J, Ferré N, Luque V, Rivero M. Feeding infant formula supplemented with the probiotic bacteria bifidobacterium longum subsp.infantis CECT7210 produce beneficial changes in gastointestinal microbial communities: a metagenomic approach. ESPGHAN Abstracts Book. JPGN. Vol. 60, Supplement 1, May 2015. PO-N-0361.